CLINICAL TRIAL: NCT06903143
Title: Piloting a Biomarker-augmented Alcohol Screening, Brief Intervention, and Referral to Treatment (SBIRT) Program Among HIV-affected Adolescents and Young Adults in Zambia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAV3113
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Alcohol
MeSH Terms: interventions — Mass Screening; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening, brief intervention, referral to treatment (SBIRT) (Experimental): Sixty AYA will be recruited from three existing HIV prevention and treatment service settings in Lusaka. These are settings where our team has both previous and current successful research studies and are real-world settings where AYA are currently receiving services. The study will be introduced to AYA during morning 'health talks' held at outpatient and ART departments as well as to AYA accessing youth friendly spaces in the three sites. Interested AYA can choose to meet with an on-site research assistant (RA). The RA will obtain informed consent and administer a brief demographics questionnaire. The RA will then conduct an alcohol screening as it would be done in the SBIRT program: the administration of the AUDIT-C screener (a 3-question brief version of the full AUDIT) and will then ask the AYA to provide a urine sample in a private bathroom. The RA will then use an EtG dipcard and after ten minutes record whether the test is positive/negative for recent alcohol consumption. The A
  Interventions: Behavioral: Screening, brief intervention, and referral to treatment (SBIRT)

INTERVENTIONS:
Behavioral: Screening, brief intervention, and referral to treatment (SBIRT) — The intervention will consist of a 30 minute alcohol brief intervention based on CETA' substance use reduction element; if warranted, referral will be made for the full CETA intervention, which consists of 6-12 weekly cognitive behavioral therapy-based sessions.

SUMMARY:
This will be a pilot study of an alcohol screening, brief intervention, and referral to treatment (SBIRT) program conducted within existing HIV prevention and treatment services for adolescents and young adults (AYA) in Lusaka, Zambia. The screening component of the program will feature both a self-report and a urine biomarker (ethyl glucuronide; EtG) to evaluate recent alcohol use. We will recruit 60 AYA to participate in the pilot. The specific aims of this pilot are to:

Specific aims:

1. Explore implementation factors of the SBIRT program within HIV prevention and treatment services through a process evaluation. We will quantitatively track the number of AYA in the SBIRT care cascade: 1) the number screened who have recent alcohol use; 2) the number of those with recent alcohol use who receive the brief intervention (BI); 3) the number of those who are referred for additional treatment; and 4) among those who are referred, the number who successfully link and complete treatment. We will collect time use data from clinic staff and counselors to estimate the time burden required for the SBIRT program. We will conduct 30 in-depth interviews with AYA three months after the screening. The sample will include adolescents who: (1) did not recently use alcohol; (2) received BI due to recent alcohol use that was low/moderate risk; and (3) were referred for treatment due to higher risk alcohol use. Interviews will focus on: (1) implementation factors (e.g., acceptability, feasibility) of the SBIRT program and (2) barriers and facilitators to the program's implementation. Focus group discussions and in-depth interviews will also be conducted with program staff (e.g., counselors, clinic staff) and other stakeholders (e.g., community leaders, policy-makers).
2. Evaluate the preliminary impact of the SBIRT program on AYA alcohol use. Among AYA who have recent alcohol use at screening, we will measure change in use at a three-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* 16-24 years of age
* Residing in Lusaka, Zambia
* Meets definition of HIV-affected as evidenced as being involved in HIV testing and treatment and Adolescent Friendly Spaces Programs at the three sites (we will not ask adolescents direct questions about HIV during screening; see Recruitment section).

Exclusion Criteria:

• Unable or unwilling to provide informed assent/consent

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) | Baseline, 3-month follow-up

SECONDARY OUTCOMES:
Ethyl glucuronide rapid dip stick | Baseline, 3-month follow=up
  EtG urine dipstick test provides positive/negative result for any alcohol use in past 2-3 days

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP